CLINICAL TRIAL: NCT00362570
Title: Phase II Trial of Continuous Dose Temozolomide in Patients With Newly Diagnosed Anaplastic Oligodendroglioma and Mixed Oligoastrocytoma
Brief Title: Temozolomide in Patients With Newly Diagnosed Anaplastic Oligodendroglioma and Mixed Oligoastrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0222
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Oligoastrocytoma, Mixed; Anaplastic Oligodendroglioma
Keywords: Newly diagnosed
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temozolomide — p.o.(by mouth), 150 mg/m2/d x days 1-7 and 15-21, given every 28 days [i.e., 7 days on/7 days off] using a standardized dosing range.
  Administration: Temozolomide will be administered on an empty stomach (i.e., 1 hour before or 2 hours after any oral intake).

SUMMARY:
Rationale:

Standard therapy for anaplastic oligodendrogliomas and mixed oligoastrocytomas includes radiation and chemotherapy. However, due to the potential long-term central nervous system toxicity from radiation, researchers speculate that it may be better to reserve radiation therapy for progressive disease. In addition, some patients with anaplastic oligodendroglioma and mixed oligoastrocytoma have unusually chemosensitive tumors. Previous research indicates that brain tumor patients with a deletion of the 1p chromosome have a higher response to the chemotherapy drug temozolomide.

DETAILED DESCRIPTION:
Temozolomide has demonstrated clinical antitumor efficacy against malignant gliomas at both relapse and initial diagnosis. This drug appears to have less adverse effects compared to other drugs used against brain tumors. Therefore, temozolomide is often better tolerated in brain tumor patients compared to other brain tumor drugs. The current study builds on previous research to test the efficacy of chemotherapy alone in patients with anaplastic oligodendroglioma and mixed oligoastrocytoma.

Purpose:

This study will evaluate response rate, or how the disease size changes in patients, and survival without disease growth, in patients with anaplastic oligodendroglioma and mixed oligoastrocytoma treated with temozolomide. Quality of life will also be assessed in this patient population treated with the study regimen.

Treatment:

Study participants will be treated with the drug temozolomide. This drug will be administered in oral pills. Temozolomide will be taken for seven consecutive days followed by seven days without the drug. This treatment schedule of seven days on temozolomide followed by seven days off will continue throughout the study. Several tests and exams will be given to closely monitor patients. MRI scans will be performed every 8 weeks to measure disease response. Temozolomide as a study drug will be given to study participants for a total of 8 week four cycles. However, treatments will be discontinued due to disease growth or unacceptable adverse events.

ELIGIBILITY:
Inclusion Criteria:

* anaplastic oligodendroglioma or mixed oligoastrocytoma
* age > 18
* Karnofsky status > 70%
* adequate bone marrow, liver and renal function

Exclusion Criteria:

* prior chemotherapy or cranial irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Determine progression free survival and response rate in patients with newly diagnosed AO and MOA of Temozolomide given every other week. | 2007-20011

SECONDARY OUTCOMES:
Assess the quality of life in this patient population using validated quality of life instruments. | 2007-2011

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Newton, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer@osu.edu